CLINICAL TRIAL: NCT04338659
Title: A Phase 1a Study Evaluating the Safety, Tolerability and Preliminary Efficacy of IBI322 in Subjects With Advanced Malignant Tumors
Brief Title: A Phase 1a Study Evaluating the Safety, Tolerability, and Efficacy of IBI322 in Subjects With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI322A102
Record Dates: First submitted 2020-03-24; First posted 2020-04-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Advanced Malignant Tumors Lymphomas
Keywords: Cancer, advanced malignancy, metastatic, solid tumor, lymphoma
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation of IBI322 (Experimental): Participants will receive escalating dose levels of IBI322 to determine maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of IBI322
  Interventions: Biological: IBI322 Recombinant anti-human CD47/PD-L1 bispecific antibody injection

INTERVENTIONS:
Biological: IBI322 Recombinant anti-human CD47/PD-L1 bispecific antibody injection — IBI322 Recombinant anti-human CD47/PD-L1 bispecific antibody injection
  Other Names: IBI322

SUMMARY:
This is a phase I study evaluating the safety, tolerability and preliminary efficacy of IBI322 in cancer subjects who failed standard treatment.

DETAILED DESCRIPTION:
A Phase 1a study evaluating the safety, tolerability and preliminary efficacy of IBI322 in subjects with advanced malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically/cytologically confirmed unresectable or metastatic solid tumors or relapsed/recurrent lymphomas for which there are no available therapies known to confer clinical benefit.
2. At least one evaluable lesion in Part A or at least one measurable lesion in Part B.
3. Male or female subject > 18 years old.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
5. Must have adequate organ function including the following.
6. Subjects with life expectancy ≥ 12 weeks.
7. Female subjects of childbearing age or male subjects whose partners are women at childbearing age, need to use 2 highly effective contraceptive measures, including one barrier method, throughout the treatment period and 6 months after the treatment period.
8. Willing to sign informed consent form and be able to comply with the study's rules and visits/related procedures.

Exclusion Criteria:

1. Previous exposure to any anti-CD47 monoclonal antibody, SIRPα antibody, or CD47/SIRPα recombinant protein.
2. Subjects participating in another interventional clinical study, except for: observational (non-interventional) clinical studies or survival follow-up phase of interventional studies.
3. Subjects who are on anticoagulants and/or require concomitant aspirin or other nonsteroids anti-inflammatory medications.
4. Subjects who have a history of blood transfusion within 2 weeks prior to screening, or the use of erythropoietin (EPO), granulocyte-colony stimulating factor (G-CSF), granulocyte-macrophage-colony stimulating factor (GM-CSF), thrombopoietin (TPO) or IL-11 therapy.
5. Subjects who received the last dose of antineoplastic therapy (chemotherapy, endocrine therapy, targeted therapy, immunotherapy or tumor embolization) within 4 weeks prior to the first dose of study drug. Subjects who received the last dose of radiotherapy within 3 weeks prior to the first dose of study drug.
6. Subjects that received immunosuppressive drugs within 7 days prior to the first dose of study drug, excluding topical, intra-nasal, or inhaled glucocorticoids or systemic glucocorticoids (i.e. equivalent to no more than 10 mg prednisone/day) or other glucocorticoids of equivalent dosage through nasal spray, inhalation or other routes.
7. Any ongoing AEs Grade 2 or higher as per NCI CTCAE v5.0 directly attributed to prior anti-tumor treatment with the exception of residual hair loss and fatigue
8. Subjects who received whole pelvic radiotherapy prior to the enrollment.
9. Subjects with known cerebrospinal metastases and other known central nervous system metastases.
10. Subjects with active or suspected autoimmune diseases or with a history of documented autoimmune disease over the past 2 years (subjects can be included in the study: vitiligo, psoriasis, alopecia or Grave's disease subjects who do not require systemic treatment within 2 years; hypothyroidism subjects who require only thyroid hormone replacement therapy, and type I diabetes subjects who require only insulin replacement therapy).
11. Known history of primary immunodeficiency.
12. Known history of active pulmonary tuberculosis.
13. Known history of allogenic organ transplantation and hematopoietic stem cell transplantation.
14. Known history of hypersensitivity to any components of the IBI322 injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | .Day 1 - Day 21
Treatment-related Adverse Events (TRAEs) | Day 1 - 90 days after last administration

SECONDARY OUTCOMES:
PK parameters | Up to 90 days post last dose
  The area under the curve (AUC)
PK parameters | Up to 90 days post last dose
  Maximum concentration (Cmax)
PK parameters | Up to 90 days post last dose
  Time at which maximum concentration (Tmax)
PK parameters | Up to 90 days post last dose
  The half-life (t1/2)
Positive rate of ADA and Nab | Up to 90 days post last dose
Positive rate of Circulating Immune Complex | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Angeles Clinic And Research Institute, Los Angeles, California
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - The University of Texas MD Anderson Cancer Center - Investigational Cancer Therapies, Houston, Texas